CLINICAL TRIAL: NCT01937338
Title: A Double Blind, Randomised, Placebo-controlled, 2-period, Cross-over Study in Healthy Volunteers to Investigate the Effects of a Single Dose of Inhaled AZD7624 on White Blood Cells and Inflammatory Markers in Induced Sputum and Blood After Oral Inhalation of 45,000 Endotoxin Units Lipopolysaccharide (LPS)
Brief Title: Study to Investigate the Effect of a Single Dose of AZD7624 on Inflammation Caused by an Endotoxin Challenge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D2550C00004
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: LPS Challenge, Neutrophils
Keywords: Healthy volunteers, Phase 1
MeSH Terms: interventions — AZD7624

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD7624 (Experimental)
  Interventions: Drug: AZD7624
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7624 — nebuliser solution; 20 mg/mL for inhalation
  Arms: AZD7624
Drug: Placebo — nebuliser solution for inhalation
  Arms: Placebo

SUMMARY:
Study to investigate the effect of a single dose of AZD7624 on inflammation caused by an endotoxin challenge.

DETAILED DESCRIPTION:
This is a double-blind, randomised, placebo controlled, 2-way cross-over study to investigate the effects of a single dose of inhaled AZD7624 on white blood cells and inflammatory markers in induced sputum and blood after oral inhalation of LPS as well as the safety, tolerability and pharmacokinetics (PK) of AZD7624 following a single inhaled dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and/or female volunteers aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture. (Healthy as determined by medical history and physical examination, laboratory parameters, and ECG performed before the first administration of the IP)
2. Female volunteers must have a negative pregnancy test at Visit 1 and on admission (Day -1 of Visit 3 and Visit 5) to the study centre, must not be lactating and must be of non childbearing potential
3. Be able to produce a minimum of 100 mg sputum (pellet weight) of good quality with total cell count (defined as total cell count <14 x 106/g, eosinophils <3%, sputum neutrophil % differential <65%, <30% squamous cell contamination and a minimum of 50% ce
4. Have normoresponsive airways with a methacholine PC20 >16 mg/mL. Screening methacholine provocation is not required if the volunteer has been tested by the centre in the past 1 year, with documented records of this testing
5. Be able to inhale from SPIRA nebuliser

Exclusion Criteria:

1. History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate
2. Any infection within the previous 4 weeks. Volunteers who get an infection between Visit 1 and admission to the centre can be rescreened
3. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or reason to expect untoward reactions to LPS and/or AZD7624
4. History of chronic respiratory disease
5. Volunteers who are vegans or have medical dietary restrictions -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Description of the pharmacodynamic Neutrophil lipopolysaccharide (LPS) response after a single dose AZD7624 in terms of % change in neutrophil differential from baseline | Sample taken at baseline visit (7-14 days before dose) and at 6h after dose day1 for each treatment. (up to 7 weeks)

SECONDARY OUTCOMES:
Description of the efficacy in terms of effect of a single dose of inhaled AZD7624 on levels of TNF-α induced sputum after oral inhalation of LPS will be evaluated compared to placebo | Sample taken at baseline visit (7-14 days before dose) and at 6h after dose day1 for each treatment. (up to 7 weeks)
Description of the safety profile in terms of Adverse events; blood pressure, heart rate and body temperature; electrocardiograms; clinical chemistry ,Creatinin kinase and myoglobin; haematology assessments, and forced expiratory volume in one second | From Screening to follow up (up to 9 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Saeed Khan, MBBS MRCP, Principal Investigator — Quintiles London, UK; Naimish Patel, Study Chair — AstraZeneca R&D Boston, United States
Locations (1):
- Research Site, London, United Kingdom